CLINICAL TRIAL: NCT02838875
Title: To Examine if the Mother's Glucose Levels and Glucose Levels in the Blood Can Predict Cord Hypoglycemia in Newborns at Risk.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0253-16-TLV
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Neonatal Hypoglycemia
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pregnant women at risk population (Experimental): women who arrived to the delivery room at Lis hospital and which the newborn is about to undergo glucose levels follow-up after birth regardless the study, because of their affiliation to the at-risk population.
  Interventions: Procedure: Blood samples

INTERVENTIONS:
Procedure: Blood samples — After birth - taking blood sample from the umbilical cord (arterial and venous) + blood sample from the patient.

SUMMARY:
Background Neonatal hypoglycemia is one of the most common metabolic disorders in neonatology. Maintaining stable levels of glucose in the transition from fetal life to life after birth is very important. Yet, except for the recognizing of at-risk populations, there are not many individual measures which can help and predict which newborns (from at-risk populations) will develop hypoglycemia and which will not.

OBJECTIVE our objective is to try to characterize by the mother's glucose levels at birth and by umbilical cord glucose levels who would be at increased risk of hypoglycemia in the hours after birth in the population that is at increased risk of this complication in advance.

DETAILED DESCRIPTION:
Background Neonatal hypoglycemia is one of the most common metabolic disorders in neonatology. Maintaining stable levels of glucose in the transition from fetal life to life after birth is very important. Yet, except for the recognizing of at-risk populations, there are not many individual measures which can help and predict which newborns (from at-risk populations) will develop hypoglycemia and which will not.

OBJECTIVE our objective is to try to characterize by the mother's glucose levels at birth and by umbilical cord glucose levels who would be at increased risk of hypoglycemia in the hours after birth in the population that is at increased risk of this complication in advance.

PATIENTS & METHODS All women who arrived to the delivery room at Lis hospital and which the newborn is about to undergo glucose levels follow-up after birth regardless the study, because his affiliation to the at-risk population including: delivery below 37th week, maternal diabetes during pregnancy and newborns in weight under percentile 10 or above percentile 90 by Dolberg graphs.

ELIGIBILITY:
Inclusion Criteria:

1. Single pregnancy
2. Vaginal or cesarean birth.
3. Births where there is an indication of neonatal hypoglycemia follow-up - one or more of the following:

   * Delivery week below 37 full weeks.
   * Maternal diabetes during pregnancy (gestational diabetes or pre-gestational).
   * Newborn under percentile 10 by Dolberg graph.
   * Newborn above percentile 90 by Dolberg graph.

Exclusion Criteria:

1. Multiple Pregnancy
2. pregnancies in which there is no indication for routine monitoring of glucose levels after birth

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Cord blood glucose levels as a predictor to newborns Hypoglycemia | 2 weeks
  Taking blood samples as a predictor to number of Hypoglycemic children.

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No